CLINICAL TRIAL: NCT00985049
Title: Whole Genome Expression of Left Ventricular Myocardium During Cardiac Surgery
Brief Title: TRANSCRIBE (Transcriptomic Analysis of Left Ventricular Gene Expression)
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Heart Association (Other); Harvard Medical School (HMS and HSDM) (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jochen Daniel Muehlschlegel, MD, Associate Professor of Anesthesia, Brigham and Women's Hospital
Other Study IDs: 2007p002323; R01HL118266 (NIH)
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, EDTA , peripheral blood leucocytes, and left ventricle myocardium are all stored in -80C frreezer at BWH.
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: The investigators hypothesize that genetic variants will alter gene expression in response to ischemia during cardiopulmonary bypass. To test this, the investigators will be taking small pieces of heart tissue from patients undergoing heart surgery before and after this period of ischemia. This will be compared to blood gene expression in blood cells and analyzed with the patients' genetic profile. This might allow us to assess the amount of inflammation that occurs when patients are on the heart-lung machine as well as examine the effects genes have on this critical time period.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than 20 years
* Undergoing aortic valve surgery with or without CABG surgery
* Receive and apical vent as part of the surgery

Exclusion Criteria:

* Will not receive an apical left ventricular vent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2009-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differential gene expression | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Jochen D. Muehlschlegel, MD, MMSc, MBA, Principal Investigator — Johns Hopkins University; Sergey Karamnov, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Heydarpour M, Ejiofor J, Gilfeather M, Stone G, Gorham J, Seidman CE, Seidman JG, Yammine M, Body SC, Aranki SF, Muehlschlegel JD. Molecular Genetics of Lidocaine-Containing Cardioplegia in the Human Heart During Cardiac Surgery. Ann Thorac Surg. 2018 Nov;106(5):1379-1387. doi: 10.1016/j.athoracsur.2018.06.016. Epub 2018 Jul 17. PMID 30028983
- [Result] Saddic LA, Nicoloro SM, Gupta OT, Czech MP, Gorham J, Shernan SK, Seidman CE, Seidman JG, Aranki SF, Body SC, Fitzgibbons TP, Muehlschlegel JD. Joint analysis of left ventricular expression and circulating plasma levels of Omentin after myocardial ischemia. Cardiovasc Diabetol. 2017 Jul 7;16(1):87. doi: 10.1186/s12933-017-0567-x. PMID 28687077
- [Result] Saddic LA, Sigurdsson MI, Chang TW, Mazaika E, Heydarpour M, Shernan SK, Seidman CE, Seidman JG, Aranki SF, Body SC, Muehlschlegel JD. The Long Noncoding RNA Landscape of the Ischemic Human Left Ventricle. Circ Cardiovasc Genet. 2017 Jan;10(1):e001534. doi: 10.1161/CIRCGENETICS.116.001534. PMID 28115490
- [Result] Sigurdsson MI, Saddic L, Heydarpour M, Chang TW, Shekar P, Aranki S, Couper GS, Shernan SK, Seidman JG, Body SC, Muehlschlegel JD. Allele-specific expression in the human heart and its application to postoperative atrial fibrillation and myocardial ischemia. Genome Med. 2016 Dec 6;8(1):127. doi: 10.1186/s13073-016-0381-1. PMID 27923400
- [Derived] Saddic LA, Chang TW, Sigurdsson MI, Heydarpour M, Raby BA, Shernan SK, Aranki SF, Body SC, Muehlschlegel JD. Integrated microRNA and mRNA responses to acute human left ventricular ischemia. Physiol Genomics. 2015 Oct;47(10):455-62. doi: 10.1152/physiolgenomics.00049.2015. Epub 2015 Jul 14. PMID 26175501